CLINICAL TRIAL: NCT06346093
Title: A Prospective, Randomised Placebo Controlled Trial of Faecal Microbiota Transplantation in Patients With Advanced Gastric Cancer
Brief Title: Fecal Microbiota Transplantation (FMT) in Patients With Advanced Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xiangyu Kong, Principle Investigator, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHEC2024-089
Record Dates: First submitted 2024-03-22; First posted 2024-04-03 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo capsules (Placebo Comparator): Placebo capsules will be administered orally three days and then every three weeks for 24 weeks. SOX and anti-PD1/PD-L1 will be intravenously infused every three weeks for 24 weeks.
  Interventions: Procedure: Placebo
- FMT capsules (Experimental): FMT capsules will be administered orally three days and then every three weeks for 24 weeks. SOX and anti-PD1/PD-L1 will be intravenously infused every three weeks for 24 weeks.
  Interventions: Procedure: Fecal Microbiota Transplantation Capsules

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation Capsules — FMT Capsules in Combination with Chemotherapy and Anti-PD1/PD-L1 Therapy
  Other Names: FMT Capsules
  Arms: FMT capsules
Procedure: Placebo — Mainly composed of starch, the appearance, shape, color, and size are exactly the same as FMT capsules
  Arms: Placebo capsules

SUMMARY:
This study is a randomized, double-blind and placebo-controlled study. The purpose of this study is to evaluate the efficacy and safety of FMT capsules combined with chemotherapy and anti-PD1/PDL1 therapy in the advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily participate in this study and provide written informed consent. Age ≥ 18 years , male or female. Pathological confirmed locally advanced, unresectable or metastatic gastric adenocarcinoma, esophagogastric junction adenocarcinoma.

Able and willing to provide tumor tissue. At least one measurable extracranial target lesion according to iRECIST. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1. Life expectancy ≥3 months.

Exclusion Criteria:

Presence of absolute contra-indications to FMT administration:Toxic megacolon;Inflammatory bowel disease;Anatomic contra-indications to colonoscopy;Colectomy Patient is currently participating and receiving other study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of this study intervention.

Currently under any form of systemic antibiotics. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (> 10 mg prednisone daily or equivalent) or any other form of immunosuppressive therapy two weeks prior to trial treatment. Patients receiving systemic steroids at physiologic doses are permitted to enroll assuming steroid dose is not above the acceptable threshold (> 10 mg prednisone daily or equivalent).

Severe anaphylactic reaction to any food (food allergies). Had a severe hypersensitivity reaction to propofol. Has serious concomitant illnesses. The eligibility can be granted by the treating investigator on individual bases.

Has HIV infection or AIDS-related illness. Has active infection of HAV, HBV or HCV. Patients with a history of Hepatitis B/C infection who have received anti-viral therapy and are disease free may be considered for enrollment after discussion with Principal Investigator.

Patient has received a live vaccine within 4 weeks prior to the first dose of treatment. Seasonal influenza vaccines or COVID-19 vaccines for injection are generally inactivated virus vaccines and are allowed.

Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Females who are pregnant or breastfeeding. Active central nervous system (CNS) metastases and/or leptomeningeal involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 6 months
  ORR is defined as the percentage of subjects who had a complete response (CR) or partial response (PR), as defined by ir-RECIST v1.1, and is based on the best response obtained.
Rate of Disease Control | up to 6 months
  Rate of Disease Control is defined as the percentage of subjects who had a complete response (CR), partial response (PR), or stable disease (SD), as defined by ir-RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 years
  The median length of time from initiation of study drug(s) disease progression as defined by RECIST v1.1, or death. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Overall Survival (OS) | up to 2 years
  The length of time (in days) from study intervention that participants remain alive.
Incidence of Adverse Events Related to Treatment | up to 6 months
  All adverse events and their relationships to study drugs and procedures will be recorded，to assess overall safety, feasibility and tolerability of treatment.
Change in the intestinal microbiome community | up to 6 months
  Mean change from baseline of bacterial species compared with 6 months post fecal microbiota transplantation (FMT).
Quality of life based on the questionnaire | up to 2 years
  The EORTC QLQ-STO22/EORTC QLQ-C30 questionnaire will be used to assess the quality of life of the participants.
Change in the immunity | up to 6 months
  Mean change from baseline of immune cells compared with 6 months post fecal microbiota transplantation (FMT).

OTHER OUTCOMES:
Marker of nutritional status | up to 2 years
  Hemoglobin is a measure of the nutritional status and are seen as markers for the catabolic state of cachectic cancer patients.
Marker of nutritional status | up to 2 years
  Creatinin is a measure of the nutritional status and is seen as markers for the catabolic state of cachectic cancer patients.
Marker of nutritional status | up to 2 years
  Albumin is a measure of the nutritional status and is seen as markers for the catabolic state of cachectic cancer patients.
Body Weight | up to 2 years
  Body Weight Change. (kilograms)
Appetite | up to 2 years
  Appetite measured by FAACT
Marker of nutritional status | up to 2 years
  C-reactief proteïne is a measure of the nutritional status and is seen as markers for the catabolic state of cachectic cancer patients.
Marker of nutritional status | up to 2 years
  Lactate dehydrogenase (LDH) is a measure of the nutritional status and is seen as markers for the catabolic state of cachectic cancer patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China